CLINICAL TRIAL: NCT00835679
Title: A Preoperative Biological Trial of Cetuximab, Dasatinib or the Combination in Colorectal Cancer Patients With Resectable Liver Metastases
Brief Title: Cetuximab and/or Dasatinib in Patients With Colorectal Cancer and Liver Metastases That Can Be Removed by Surgery
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NCI-2013-00014; NCI-2013-00014 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VU-VICC-GI-0838; 8069; P30CA068485 (NIH); 081338; VICC GI 0838 (Other: Vanderbilt-Ingram Cancer Center); 8069 (Other: CTEP)
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2013-01

CONDITIONS: Liver Metastases; Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Dasatinib

ARMS (4):
- Cohort A (no systemic neoadjuvant therapy) (Experimental): Patients receive no systemic neoadjuvant therapy between enrollment and the time of definitive surgical resection of liver metastases. Liver biopsies were performed at surgery since this cohort received no systemic therapy.
  Interventions: Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis
- Cohort B (cetuximab) (Experimental): Patients receive 400 mg/m^2 cetuximab IV over 120 minutes on day 1 and 250 mg/m^2 cetuximab IV over 60-120 minutes on day 8. Definitive surgical resection of liver metastases will take place on day 15.
  Interventions: Biological: cetuximab; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis
- Cohort C (dasatinib) (Experimental): Patients receive dasatinib 100 mg orally once daily on days 1-14. Definitive surgical resection of liver metastases will take place on day 15.
  Interventions: Drug: dasatinib; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis
- Cohort D (cetuximab, dasatinib) (Experimental): Patients receive 400 mg/m^2 cetuximab IV over 120 minutes on day 1 and 250 mg/m^2 cetuximab IV over 60-120 minutes on day 8 AND dasatinib 100 mg orally once daily on days 1-14. Definitive surgical resection of liver metastases will take place on day 15.
  Interventions: Biological: cetuximab; Drug: dasatinib; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
  Arms: Cohort B (cetuximab); Cohort D (cetuximab, dasatinib)
Drug: dasatinib — Given orally
  Other Names: BMS-354825; Sprycel
  Arms: Cohort C (dasatinib); Cohort D (cetuximab, dasatinib)
Procedure: therapeutic conventional surgery — Undergo surgery
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase 0 trial is studying whether 2 weeks of cetuximab and dasatinib will change tumor cells in patients with colorectal cancer and liver metastases that can be removed by surgery. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the biological effects of cetuximab, dasatinib, or the combination on epidermal growth factor receptor (EGFR)- and Src-signaling pathways in resected colorectal cancer liver metastases.

OUTLINE: This is a multicenter study. Patients are initially enrolled in cohort A. Once cohort A is completed, additional patients are enrolled and randomized to treatment in either cohorts B or C. If a significant biological effect is seen in cohorts B or C, additional patients are enrolled in cohort D.

COHORT A: Patients receive no systemic neoadjuvant therapy between enrollment and the time of definitive surgical resection of liver metastases. Liver biopsies were performed at surgery since this cohort received no systemic therapy.

COHORT B: Patients receive 400 mg/m2 cetuximab intravenously (IV) over 120 minutes on day 1 and 250 mg/m^2 cetuximab IV over 60-120 minutes on day 8. Definitive surgical resection of liver metastases will take place on day 15.

COHORT C: Patients receive dasatinib 100 mg orally once daily on days 1-14. Definitive surgical resection of liver metastases will take place on day 15.

COHORT D: Patients receive 400 mg/m^2 cetuximab IV over 120 minutes on day 1 and 250 mg/m^2 cetuximab IV over 60-120 minutes on day 8 AND dasatinib 100 mg orally once daily on days 1-14. Definitive surgical resection of liver metastases will take place on day 15.

Patients undergo tumor tissue (from initial liver tumor biopsies and liver resection samples), serum, and peripheral blood mononuclear cell sample collection periodically for biomarker analysis via immunohistochemistry (IHC).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed adenocarcinoma arising from the large intestine that has metastasized to the liver; liver metastases may be synchronous or metachronous
* The liver metastases must be considered surgically resectable prior to the initiation of study drugs
* Prior chemotherapy or chemoradiotherapy for colorectal cancer is allowed provided that toxicities from prior therapy have resolved to Grade 1 or less; no prior anti-EGFR or anti-Src therapy is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Absolute neutrophil count >= 1.5 x 10^9/L
* Hemoglobin ≥ 9.0 Gm/dL
* Platelets >= 100 x 10^9/L
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine transaminase (ALT)(serum glutamic pyruvic transaminase [SGPT]) =< 5 x institutional upper limit of normal
* Creatinine =< 1.5 institutional ULN
* Women must have a negative pregnancy test; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Although KRAS status will be evaluated in the tumor, wild type KRAS status is not an eligibility criterion

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cetuximab or dasatinib
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cetuximab or dasatinib, breastfeeding should be discontinued if the mother is treated with cetuximab or dasatinib
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with cetuximab or dasatinib; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients on potent CYP3A4 inducers and inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Chan, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to accrual from December 2009 to August 2011.
Pre-assignment Details: Eleven patients consented, with two ineligible. The study closed prematurely due to slow accrual.
Groups:
- No Treatment Cohort A: Patients receive no systemic neoadjuvant therapy between enrollment and the time of definitive surgical resection of liver metastases. Liver biopsies were performed at surgery since this cohort received no systemic therapy.
- Cetuximab Cohort B: Patients receive 400 mg/m2 cetuximab intravenously (IV) over 120 minutes on day 1 and 250 mg/m2 cetuximab IV over 60-120 minutes on day 8. Definitive surgical resection of liver metastases will take place on day 15
- Dasatinib Cohort C: Patients receive dasatinib 100 mg orally once daily on days 1-14.Definitive surgical resection of liver metastases will take place on day 15
- Cetuximab + Dasatiib Cohort D: Patients receive 400 mg/m2 cetuximab intravenously (IV) over 120 minutes on day 1 and 250 mg/m2 cetuximab IV over 60-120 minutes on day 8 AND dasatinib 100 mg orally once daily on days 1-14. Definitive surgical resection of liver metastases will take place on day 15
Period: Overall Study
Arm/Group | No Treatment Cohort A | Cetuximab Cohort B | Dasatinib Cohort C | Cetuximab + Dasatiib Cohort D
Started | 9 | 0 (This study closed prematurely, thus no patients went on Cohort B, C or D.) | 0 | 0
Completed | 8 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Treatment Cohort A | Cetuximab Cohort B | Dasatinib Cohort C | Cetuximab + Dasatiib Cohort D | Total
Number analyzed (Participants) | 9 | 0 | 0 | 0 | 9
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  |  |  | 0
  Between 18 and 65 years | 7 |  |  |  | 7
  >=65 years | 2 |  |  |  | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (1) |  |  |  | 58 (1)
Gender [Number; unit: participants]
  Female | 5 |  |  |  | 5
  Male | 4 |  |  |  | 4
Region of Enrollment [Number; unit: participants]
  United States | 9 |  |  |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Patients With a Biologic Response
Description: Patients who experienced a pre-to-post treatment reduction of at least 1 scoring level from baseline on preoperative-day 15 in at least 1 biomarker of the pathway being inhibited: epidermal growth factor (EGFR) for Cohort B, sarcoma (Src) for Cohort C, and both EGFR and Src for Cohort D. Blood for these biomarkers will be taken on day of baseline and pre-operatively on day 15. Determined by 0-4-scale scoring with score determined by percentage of tumor cells positively stained for pathway in question: minimum 0 (0%), 1 (1-24%), 2 (25-49%), 3 (50-74%), and maximum 4 (75-100%).
Time Frame: on baseline and preoperatively on day of surgery (day 15)
Population: No patients accrued to Cohorts B, C, and D, who were to receive the study drugs. Nine patients were accrued in Cohort A; these patients received no study drugs and were to determine normal levels of selected biomarkers. No biomarkers were determined; no data available. This study was closed prematurely due to slow accrual.
Groups:
- Cetuximab +Dasatinib Cohort D: Patients receive 400 mg/m2 cetuximab intravenously (IV) over 120 minutes on day 1 and 250 mg/m2 cetuximab IV over 60-120 minutes on day 8 AND dasatinib 100 mg orally once daily on days 1-14. Definitive surgical resection of liver metastases will take place on day 15
Arm/Group | No Treatment Cohort A | Cetuximab Cohort B | Dasatinib Cohort C | Cetuximab +Dasatinib Cohort D
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Patients With Reduction of Biomarkers in Tumor Tissue
Description: Patients with pre-to-post treatment reduction at least 1 scoring level from baseline on preoperative-day 15 in at least 1 biomarker: total & phi-EGFR, phi-MAPK, phi-Akt, Ki67, phi-FAK, phi-paxillin, phi-Src, capase 3. Determined by 0-4-scale scoring with score determined by percentage of tumor cells positively stained for biomarker in question: minimum 0 (0%), 1 (1-24%), 2 (25-49%), 3 (50-74%), and maximum 4 (75-100%)
Time Frame: study entry to day 15
Population: as for outcome 1
Arm/Group | No Treatment Cohort A | Cetuximab Cohort B | Dasatinib Cohort C | Cetuximab + Dasatiib Cohort D
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Patients With the Given Severity of Adverse Event Within a Specified Duration
Description: Number of patients with each grade of adverse event (AE) during the specified timeframe using the Common Terminology Criteria for AEs guide, grades 1-5 with one being mild, five is death.
Time Frame: weekly to day 15, and at followup on day 30
Population: No patients accrued to Cohorts B, C, and D, which were to receive the study drugs. Nine patients were accrued in Cohort A; these patients received no study drugs and were to determine normal levels of selected biomarkers. No patients were accrued to Cohorts B, C, D. This study was closed prematurely due to slow accrual.
Groups:
- No Treatment Cohort A: Patients receive no systemic neoadjuvant therapy between enrollment and definitive surgical resection of liver metastases. Liver biopsies were performed at surgery since this cohort received no systemic therapy.
- Dasatinib Cohort C: Patients receive dasatinib 100 mg orally once daily on days 1-14.Definitive surgical resection of liver metastases will take place on day 15 1-14.
- Cetuximab + Dasatinib Cohort D: Patients receive 400 mg/m2 cetuximab intravenously (IV) over 120 minutes on day 1 and 250 mg/m2 cetuximab IV over 60-120 minutes on day 8 AND dasatinib 100 mg orally once daily on days 1-14. Definitive surgical resection of liver metastases will take place on day 15
Arm/Group | No Treatment Cohort A | Cetuximab Cohort B | Dasatinib Cohort C | Cetuximab + Dasatinib Cohort D
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Patients With the Given Severity of Post-operative Complications Within the Specified Duration
Time Frame: From day 15 (day of surgery) to 30 days after surgery
Population: No patients accrued to Cohorts B, C, and D, which were to receive the study drugs. Nine patients were accrued in Cohort A; these patients received no study drugs and were to determine normal levels of selected biomarkers.No patients received any study drugs. This study was closed prematurely due to slow accrual.
Arm/Group | No Treatment Cohort A | Cetuximab Cohort B | Dasatinib Cohort C | Cetuximab + Dasatiib Cohort D
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | No Treatment Cohort A | Cetuximab Cohort B | Dasatinib Cohort C | Cetuximab + Dasatiib Cohort D
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/9 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to study design and slow accrual, no drug was received, no biomarkers were determined and no data obtained. "0" data is entered in the outcomes measures database as suggested by CT.gov previously. Detailed explanations are given.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less